CLINICAL TRIAL: NCT00811226
Title: Prospective, Multicentric, Open Clinic Essay to Evaluate the Use of OLMETEC® (Olmesartan Medoxomile) and OLMETEC PLUS® (Olmesartan Medoxomile Hydrochlorothiazide) in Stade I and II, According to JNC VII
Brief Title: Assessment of the Effectiveness of OLMETEC® and OLMETEC PLUS® for Treatment of Hypertension in Stage I and II Patients (Study P05254)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Schering-Plough (Industry)
Responsible Party: Head, Clinical Trials Registry & Results Disclosure Group, Schering-Plough
Other Study IDs: P05254
Record Dates: First submitted 2008-07-25; First posted 2008-12-18 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Hypertension
Keywords: Hypertension Stage I; Hypertension Stage II
MeSH Terms: conditions — Hypertension | interventions — Hydrochlorothiazide; Olmesartan Medoxomil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients with arterial hypertension Stade I or Stade II
  Interventions: Drug: olmesartan medoxomile alone or combined with hydrochlorothiazide,

INTERVENTIONS:
Drug: olmesartan medoxomile alone or combined with hydrochlorothiazide, — olmesartan medoxomile 20mg/daily or 40mg/daily; olmesartan medoxomile 20mg plus 12.5 mg of hydrochlorothiazide daily; olmesartan medoxomile 40mg plus 12.5 mg of hydrochlorothiazide daily
  Other Names: SCH 900332; OLMETEC®; OLMETEC PLUS ®

SUMMARY:
The purpose of this study is to determine the efficiency of Olmesartan medoxomile (OLMETEC®) alone or in combination with hydrochlorothiazide (OLMETEC PLUS®) in the reduction of arterial blood pressure in patients with light to moderate hypertension, and to evaluate the percentage of patients that reach treatment goals using this antihypertensive regimen.

DETAILED DESCRIPTION:
α= 0.05. α's Z=1.96 β= 80%. β's Z=0.84 Estimated proportion of subjects to achieve optimal control of arterial hypertension= 83.2%

450 subjects are expected to be enrolled in the study of which 40 subjects will be enrolled in Venezuela.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 years of age or older
* Essential arterial hypertension Stade I and II according to JNC VII
* Signature of Informed Consent

Exclusion Criteria:

* Secondary arterial hypertension
* Pregnant woman or during lactancy
* Recent cardiovascular disease, as heart attack, unstable angina, or procedures of coronary revascularization on the previous six months.
* Acute Coronary Failure Syndrome on the previous six months.
* Chronic Ischemic Cardiopathy Treatment.
* Cerebral Vascular Disease on the previous six months.
* Alcoholism Story or use of drugs on the two previous years.
* Hepatic Disease Story
* Chronic Renal Failure defined by a serumal creatinine higher than 2mg/dl
* Albuminuria higher than 1gr.
* Known Allergy to blockers of angiotensine II receptors.
* Neoplasmic Malignant Disease included leukemia and the lymphoma (Skin basocellular cancer is not included)
* Auto Immune Disorders as systemic erythematosus lupus.
* Non attachment to medical treatments history.
* Patients sharing some clinical investigation essay on the last 3 months.
* Congestive heart failure under previous treatment with ECA inhibitors.
* Allergy to thiazidic diuretics.
* Angioedema History
* Use of drugs that affect potassium secretion, as diuretic savers of potassium, angiotensine enzyme inhibitor, betablockers, non-steroid anti-inflammatory drugs.
* Potassium consumption orally

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in Venezuela with arterial hypertension Stade I or Stade II
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2007-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the efficiency of Olmesartan medoxomile (OLMETEC®) alone, or in combination with hydrochlorothiazide (OLMETEC PLUS®) in decreasing diastolic pressure | basal registry and on follow-up visits in weeks 4, 8, 12, and 16

SECONDARY OUTCOMES:
Evaluation of the efficiency of Olmesartan medoxomile (OLMETEC®) alone, or in combination with hydrochlorothiazide (OLMETEC PLUS®) in decreasing systolic pressure | basal registry and on follow-up visits in weeks 4, 8, 12, and 16
Evaluation of the percentage of patients (including diabetics and those with renal disease) that achieve arterial blood pressure treatment goals with Olmesartan medoxomile (OLMETEC®) alone, or in combination with hydrochlorothiazide (OLMETEC PLUS®) | basal registry and on follow-up visits in weeks 4, 8, 12, and 16